CLINICAL TRIAL: NCT04239443
Title: Peripheral Circulating Blood Tumor Cells (CTC) Detection and CTC-based PD-L1 Antibody Immunofluorescence Detection to PD-1 Monoclonal Antibody SHR-1210 and Apatinib in Second-line and Back-line Treatment of Advanced NSCLC, Soft Tissue Sarcoma, Uterine Cancer Clinical Research
Brief Title: Clinical Study of PD-1 Monoclonal Antibody SHR-1210 and Apatinib in Advanced NSCLC, Soft Tissue Sarcoma, and Uterine Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCHIIT001
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Advanced Non Small Cell Lung Cancer; Uterine Cancer; Soft Tissue Sarcoma
Keywords: immunotherapy; PD-1 checkpoint inhibitor; circulating blood tumor cells (CTC)
MeSH Terms: conditions — Uterine Neoplasms; Sarcoma | interventions — Immune Checkpoint Inhibitors; camrelizumab; apatinib

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in our study. NSCLC participants will be given intravenous administration of SHR-1210 (200mg/2w) and oral of Apatinib (250mg/d) , soft tissue sarcoma will be given intravenous administration of SHR-1210 (200mg/3w) and oral of Apatinib (500mg/d), and uterine cancer will be given intravenous administration of SHR-1210 (200mg/3w) and oral of Apatinib (250mg/d).
  Treatments will be administrated until disease progression, death, or unacceptable toxicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1210 and Apatinib (Experimental): NSCLC participants will be given intravenous administration of SHR-1210 (200mg/2w) and oral of Apatinib (250mg/d) , soft tissue sarcoma will be given intravenous administration of SHR-1210 (200mg/3w) and oral of Apatinib (500mg/d), and uterine cancer will be given intravenous administration of SHR-1210 (200mg/3w) and oral of Apatinib (250mg/d).
  The duration of treatment will till the disease progression, death, or unacceptable toxicity show up.
  Interventions: Drug: PD-1 inhibitor; Drug: Apatinib

INTERVENTIONS:
Drug: PD-1 inhibitor — Intravenous administration of SHR1210 (200mg/2weeks or 200mg/3weeks)
  Other Names: Camrelizumab
Drug: Apatinib — NSCLC and Uterine cancer will be given oral of Apatinib (250mg/d), soft tissue sarcoma will be given oral of Apatinib (500mg/d).

SUMMARY:
In this one-arm study, histologically or cytologically confirmed advanced NSCLC, uterine malignancies, and soft tissue sarcoma will be enrolled to investigate the efficacy and safety of PD-1 monoclonal antibody SHR-1210 and apatinib, at the same time, peripheral circulating blood tumor cells (CTC) detection and CTC-based PD-L1 antibody immunofluorescence detection will be performed.

DETAILED DESCRIPTION:
Primary outcome:

1. Analysis of baseline levels of CTC and CTC PD-L1 and prognosis efficacy of patients: Objective remission rate (ORR), progression free survival (PFS), overall survival (OS);
2. Dynamic monitoring of CTC and CTC PD-L1 at baseline before treatment, after two cycles of treatment, and as the disease progresses.
3. Consistency analysis of PD-L1 and CTC PD-L1 expression in tissue specimens.

Secondary outcome:

Duration of response(DOR), Disease control rate(DCR), Safety of the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years, both men and women (Uterine cancer limited to women);
2. NSCLC: Pathologically confirmed advanced (IIIB, stage IV) NSCLC with at least 1 measurable lesion that meets the RECIST v1.1 standard without local treatment, of which stage IIIb patients are incapable, unsuitable for surgery or radical radiotherapy, NSCLC patients have failed at least the first-line standard treatment or refused to receive standard treatment, or chemotherapy intolerance, Among them, patients with sensitive gene mutations must fail after TKI treatment (patients who have failed first-line or second-line treatment may participate in this study), Patients with EGFR and ALK mutations must undergo EGFR and ALK inhibitor treatment failure and EGFR T790M mutation negative, for EGFR T790M-positive patients, third-generation EGFR TKI treatment fails.
3. Soft tissue sarcoma: Patients with distant metastasis or locally advanced disease who have previously failed chemotherapy or sensitive recurrence or metastasis to soft tissue sarcoma. Subjects who have judged by the investigator to be unsuitable for surgical treatment (including amputation) of soft tissue sarcomas (diagnosed pathologically or cytologically, but excluding gastrointestinal stromal tumors, chondrocyte-bone tumors, embryonic/acinar rhabdomyosarcoma, Juventus Sarcoma, extensive distant metastatic soft tissue tumors such as keloid cutaneous fibrosarcoma and inflammatory myofibroblastic sarcoma, malignant peripheral nerve sheath tumor, keloid cutaneous fibrosarcoma, inflammatory myofibroblastic sarcoma, malignant interstitial Dermatoma) (priority consideration: synovial sarcoma, undifferentiated multiline sarcoma, dedifferentiated liposarcoma), and measurable lesions that meet the RECIST 1.1 standard.
4. Uterine cancer: Pathologically confirmed uterine cancer, including cervical cancer (squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma), endometrial cancer, and uterine sarcoma, at least one measurable lesion that meets RECIST 1.1 criteria, recurrence/Persons with persistent cervical cancer, endometrial cancer, and uterine sarcoma cannot be cured by surgery and/or radiotherapy, have received at least a first-line treatment for advanced (stage IVB), recurrent/persistent cervical cancer, endometrial cancer, uterine sarcoma Systemic chemotherapy patients (qualified to participate in this study after the progress of first-line chemotherapy).
5. All acute toxicity caused by previous antitumor treatments were alleviated to level 0-1 (according to NCI CTCAE version 4.03) or to the level specified by the enrollment/ exclusion criteria 1 day before the first dose except for subjects whose toxicity does not pose a safety risk);
6. Able to provide tumor samples (at least 20 unstained tumor samples or fresh tissue specimens embedded in formalin-fixed paraffin within six months, 4ml of peripheral blood samples before treatment and each effect evaluation);
7. ECOG score: 0-1, patients with soft tissue sarcoma amputation can be relaxed to 2 points;
8. Expected survival ≥ 12 weeks;
9. The function of important organs meets the following requirements (excluding the use of any blood components and cell growth factors during screening);

   1. Absolute neutrophil count ≥1.5 × 109 / L;
   2. platelets ≥100 × 109/L;
   3. Hemoglobin ≥9g/dL;
   4. serum albumin ≥3g/dL;
   5. total bilirubin ≤ 1.5ULN;
   6. ALT and AST ≤1.5ULN;
   7. AKP ≤ 2.5ULN;
   8. Serum creatinine ≤ 1.5ULN or creatinine clearance ≥ 60mL/min;
10. Non-surgical sterilization female patients;
11. Participants volunteered to participate in the study, signed informed consent, good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Participants who had any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis , Hyperthyroidism, decreased thyroid function; subjects with vitiligo or childhood asthma has completely resolved, adults can be included without any intervention; subjects with bronchodilators for medical intervention can not be included in asthma;
2. Participants who were treated with immunosuppressive agents, or systemic or absorbable local hormones for immunosuppressive purposes (dose>10mg/day, prednisone or other curative hormones), and continued to use it within 2 weeks before enrollment;
3. Excessive allergic reactions to other monoclonal antibodies;
4. Participants who had clinical symptoms of central nervous system metastases (such as brain edema, require hormonal intervention, or progress of brain metastases). Participants who had previously received brain or meningeal metastasis treatment, such as clinical stability (MRI) that has been maintained for at least 1 month, and have stopped systemic hormonal therapy (dose> 10 mg / day prednisone or other therapeutic hormone) can be included;
5. Imaging (CT or MRI) showed that the tumor invades or demarcates large blood vessels.
6. Imaging (CT or MRI) showed obvious hollow or necrotic tumors in the lungs; those with marginal adenocarcinoma with cavities can be considered after discussion with the clinician.
7. Participants who had high blood pressure and cannot be well controlled with antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90 mmHg).
8. Participants who had poorly controlled clinical symptoms or diseases of the heart, such as: (1) heart failure above NYHA 2 (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular Sexual arrhythmias require treatment or intervention.
9. Participants who had abnormal blood coagulation (PT> 16s, APTT> 43s, TT> 21s, Fbg <2g / L), bleeding tendency or receiving thrombolytic or anticoagulation；
10. Urine routine indicates urinary protein ≥ ++, or confirms that 24-hour urine protein is ≥1.0 g；
11. Participants who previously received radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy. After treatment is completed (last dose), subjects less than 4 weeks before study medication (or 5 drug half-life, whichever is longer) Patients who did not recover from adverse events (excluding hair loss) from previous treatment to ≤CTCAE 1 degree；
12. Clinically ascites or pleural effusion requiring therapeutic puncture or drainage；
13. Participants who had obvious cough blood in the first 2 months of randomization, or a day with hemoptysis of half teaspoon (2.5ml) or more；
14. Participants who had clinically significant bleeding symptoms or have a clear bleeding tendency within the first 3 months of randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood at baseline and above, or have vasculitis；
15. Participants who had arterial/venous thrombotic events such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism occurred within the first 6 months；
16. Participants who had known hereditary or acquired bleeding and thrombotic tendency (eg hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.)；
17. Participants who had an active infection or an unexplained fever during the screening period before the first dose> 38.5 degrees;
18. Patients with past and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of lung function, etc;
19. Participants who had congenital or acquired immune deficiency (such as HIV-infected persons), or positive for syphilis spiral antibodies, or active hepatitis (HBV reference: HBsAg positive, and HBV DNA detection exceeds the upper limit of normal values; (And the HCV virus titer detection value exceeds the upper limit of normal value);
20. Participants who have used other drugs in clinical trials within 4 weeks before the first use;
21. Participants has previous or concurrent other malignancies (except cured skin basal cell carcinoma and cervical carcinoma in situ);
22. Participants may receive other systemic anti-tumor treatments during the study;
23. Participants with bone metastases who had received palliative radiation therapy within 4 weeks before participating in the study;
24. Participants who have previously received other PD-1 antibody treatments or other immunotherapy against PD-1/PD-L1 or VEGFR single-target/multi-target inhibitors, such as Sunitinib, Sorafeni, Bevacizumab, Anlotinib, Famitinib, Apatinib, and Reginafinib (in advanced NSCLC, there is no need to exclude previous VEGFR single / multitarget inhibitor Patients treated, but need to be discontinued for more than 4 weeks);
25. Live vaccine may be given less than 4 weeks before study medication or possibly during the study;
26. According to the researcher's judgment, Participants has other factors that may lead to the termination of the study. Serious diseases (including mental illness) require combined treatment. There are serious laboratory abnormalities, accompanied by family or social factors. To the safety of the subject, or the collection of information and samples;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Progression free survival (PFS) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Overall survival (OS) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
The number of Circulating Tumor Cell (CTC) | 2 years
Analysis of PD-L1 expression on Circulating Tumor Cell (CTC) and tumor tissue | 2 years

SECONDARY OUTCOMES:
Duration of response(DOR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Disease control rate(DCR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, Principal Investigator — Hunan Cancer Hospital; Kunyan Li, Principal Investigator — Hunan Cancer Hospital; Jing Wang, Principal Investigator — Hunan Cancer Hospital; Gang Huang, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author of published work.